CLINICAL TRIAL: NCT00575926
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study of the Clinical Effects of Ganoderma Lucidum (Ling Zhi) in Children With Cancer
Brief Title: Lingzhi for Cancer Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Dr. Matthew Ming-kong Shing, MBBS, FRCP, Department of Pediatrics, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCFGrants2000.MKS
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Pediatric Cancers
Keywords: Randomized controlled trial; Lingzhi; Immune functions; Quality of life; Survival

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Lingzhi extract (Active Comparator): Oral 300mg capsules containing Lingzhi extract (4 to 6 capsules per day as dosed by patients' age)
  Interventions: Drug: LingZhi capsule
- B: Placebo (Placebo Comparator): Starch with same appearance and taste as LingZhi
  Interventions: Drug: LingZhi capsule

INTERVENTIONS:
Drug: LingZhi capsule — LingZhi or Placebo 300 mg x 4 or 300 mg x 6 capsules daily according to age group
  Other Names: Ganoderma lucidum

SUMMARY:
Ganoderma lucidum (Lingzhi) is a Traditional Chinese Medicine which is widely used as a means to 'strengthen immunity' among patients with cancers. However, there is no published randomized controlled clinical trial on its efficacy and safety despite the many in vitro studies on its anti-viral, anti-oxidative, anti-tumour, radioprotective, hepato-protective and immunomodulatory effects. This study was a randomized, double-blind, placebo-controlled, parallel clinical trial that investigated the benefits and safety of Ganoderma lucidum (Lingzhi) in treating children with cancers. Patients were randomized to receive identical capsules of either Lingzhi or placebo for six months. The primary outcome was the general Paediatric Quality of Life score. Secondary outcomes included immune functions, infection-related morbidities, complete blood counts and serum biochemistry, and overall and event-free survival.

DETAILED DESCRIPTION:
Alternative and complementary medicine are widely used in treating children with cancers. A population-based survey in British Columbia revealed that they were used by 42% of the respondents. Among Chinese in Hong Kong, Traditional Chinese Medicine (TCM) is also widely practiced. Some 60% of the population had consulted TCM practitioners at one time or another. TCM use could be dated back to more than five thousand years ago, and written records were available for over two thousand years. TCM is considered to be an integral part of the Chinese culture. In our experience, TCM is believed to be commonly used to 'strengthen immunity and promote health' among local children with cancers, despite the lack of well-designed study to prove its usefulness. Ganoderma lucidum (Ling Zhi) is a mushroom long-used in China for a broad range of disorders. Its use is common in the general population and among both adults and children with a wide range of malignancies. However, there is no randomized controlled trial to support its clinical efficacy and safety. Therefore, we conducted this clinical trial of Ganoderma lucidum (Ling Zhi) among Hong Kong children with cancers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 2-18 years
* Acute lymphoblastic leukaemia who completed induction chemotherapy and pending maintenance chemotherapy treatment
* Solid tumours completed chemotherapy
* Aute myeloid leukaemia who completed induction and consolidation chemotherapy treatment
* All patients and their parents signed informed written consent

Exclusion Criteria:

* Relapsed cancer patients
* Received Traditional Chinese Medicine (TCM) treatment within preceding one month
* Could not swallow capsules
* Syndromal disorders (e.g. Down syndrome)
* History of hypersensitivity reaction to Lingzhi or any TCM
* Significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, cardiovascular or allergic diseases
* In the judgement of investigators were unable to comply with study protocol requirements

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2002-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Generic and cancer-specific Pediatric Quality-of-Life assessment | 1 year

SECONDARY OUTCOMES:
Cellular immune functions; blood counts and biochemistry for patient safety; infection-related morbidities; overall and event-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew MK Shing, MBBS, FRCP, Principal Investigator — Department of Pediatrics, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Department of Pediatrics and Adolescent Medicine, Princess Margaret Hospital, Hong Kong
  - Department of Pediatrics, Queen Elizabeth Hospital, Hong Kong
  - Department of Pediatrics, The Chinese University of Hong Kong, Hong Kong